CLINICAL TRIAL: NCT01608503
Title: The Effect of Lung Deflation on the Position of the Pleura in Mechanically Ventilated Infants During Subclavian Vein Cannulation: an Ultrasound Study
Brief Title: Lung Deflation in Pediatric Subclavian Vein Catheterization
Acronym: SCVLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: SVCLungDown
Record Dates: First submitted 2012-05-26; First posted 2012-05-31 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Pediatric Subclavian Vein Catheterization
Keywords: subclavian vein; ultrasound; distance between the subclavian vein and the lung

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- respiration cycle (Experimental): lung inflation and deflation
  Interventions: Procedure: lung deflation; Procedure: lung inflation

INTERVENTIONS:
Procedure: lung deflation — lung was deflated during respiration cycle
Procedure: lung inflation — lung was inflated during respiratory cycle

SUMMARY:
The subclavian vein (SCV) is a preferred site for placement of central venous catheter. However, pneumothorax is a major concern during subclavian venous catheterization. Lung deflation, by decreasing lung volume, may reduce the risk of pneumothorax by increasing the distance between the pleura and the SCV. The investigators evaluated the effect of lung deflation on the relative position between the pleura and the line of the imaginary needle pathway during supraclavicular and infraclavicular approach to the subclavian vein (SCV) using ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who were scheduled for elective operation under general anesthesia
* Neonates (0 ~ 1 mo), Infants (1 mo ~ 1 yr)

Exclusion Criteria:

* Structural anomalies of the chest wall
* History of lung and chest wall operations
* Prior central venous catheterization
* Upper respiratory tract infection, or pneumonia within 2 weeks

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The distance between the pleura and the line of the imaginary needle pathway (DPI) | Within 5 minutes
  The ultra-sonography probe was adjusted to obtain an image containing the long-axis cross section of SCV, the pleura, the clavicle, and the first rib. Images were recorded by the same physician during whole respiratory cycle with the probe held in the identical position.
  Imaginary lines for supraclavicular and infraclavicular approach were drawn, and distances from the pleura were measured.
  If the pleura touched the INP, the distance was recorded as positive value. If the pleura did not touch the INP, the distance was recorded as negative value.

SECONDARY OUTCOMES:
The incidence of pleural movement over the imaginary needle pathway | Within 5 minutes
  If the pleura touched the imaginary needle pathway, the incidence was checked.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea